CLINICAL TRIAL: NCT01578915
Title: A Case Control Study of Women With Multiple Sexual Partners Attending the Jefferson County Department of Health Sexually Transmitted Diseases Clinic
Brief Title: A Case Control Study of Women With Multiple Sexual Partners
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Christina Muzny, Assistant Professor of Medicine, University of Alabama at Birmingham
Other Study IDs: High Risk Women
Record Dates: First submitted 2012-03-04; First posted 2012-04-17 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Women with 4 or more sexual partners during the past year
- Controls: Women with only one sexual partner during the past year

SUMMARY:
Both population based surveys and more focused research studies indicate that increased numbers of sexual partners and partner concurrency contribute to increased risk for acquisition of sexually transmitted infection (STI), including HIV infection. However, unlike for men, both national and sub-population-based studies consistently find that the great majority of women with or without STIs report only 1-2 sex partners in the preceding year and that a minority of women acknowledge > 3 sex partners over the same period, suggesting that this relatively small proportion of women with higher numbers of sex partners play a disproportionate role in sustaining community STI rates. Despite these observations, surprisingly little is known about women with increased numbers of sexual partners, the factors which contribute to increased partner number, and the potential for those factors to be intervened upon to reduce risk for STI. The implications of these facts for STI/HIV prevention efforts are profound. For instance, interventions that include the implication that target audiences have multiple sex partners might be dismissed as irrelevant by those with single partners. Conversely, interventions targeting women with multiple sex partners may be based on assumptions derived from data which, while representative of the general target audience, may not reflect relevant circumstances for the subset of women with higher numbers of partners.

This study will begin to generate data that will provide critical information on this topic and help inform future development of STI/HIV interventions tailored to womens' individual circumstances and contexts. The investigators hypothesize that women with 4 or more sexual partners during the past year will report higher rates of depression and substance abuse (alcohol and drugs), higher rates of intimate partner violence, less social support, more non-vaginal sex, more same-sex contacts, and higher rates of STIs than women reporting only one sexual partner during the past year.

DETAILED DESCRIPTION:
The objectives of this protocol are: (1) To delineate factors that are important modifiable predictors of sexually transmitted infection (STI) risk in the context of increased numbers of sexual partners, comparing those participants with one sexual partner to those with 4 or more sexual partners during the past year. (2) To define the prevalence of infection with Chlamydia, gonorrhea, trichomoniasis, syphilis, genital herpes, and HIV in women reporting one sexual partner in the past year compared to women reporting 4 or more sexual partners during the past year.

ELIGIBILITY:
Inclusion Criteria:

* female,
* age 16 years or older,
* report of either one sexual partner during the past year or 4 or more sexual partners in the past year,
* able to provide written informed consent

Exclusion Criteria:

* Drug and/or alcohol intoxication at the time of enrollment,
* exhibition of any type of disruptive or unsafe behavior that would not be conducive to participating in this study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women presenting to the Jefferson County Department of Health Sexually Transmitted Diseases Clinic
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
STI diagnosis | Day of enrollment

SECONDARY OUTCOMES:
Sexual risk behaviors | Up to 3 months prior to enrollment
Substance use (alcohol and drugs) | Up to 30 days prior to enrollment
History of intimate partner violence | At any time prior to enrollment
Depression | Up to 7 days prior to enrollment
Social support | Up to 30 days prior to enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Muzny, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Jefferson County Department of Health, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Wagoner NJ, Harbison HS, Drewry J, Turnipseed E, Hook EW 3rd. Characteristics of women reporting multiple recent sex partners presenting to a sexually transmitted disease clinic for care. Sex Transm Dis. 2011 Mar;38(3):210-5. doi: 10.1097/OLQ.0b013e3181f6fe42. PMID 20966829
- [Background] Santelli JS, Brener ND, Lowry R, Bhatt A, Zabin LS. Multiple sexual partners among U.S. adolescents and young adults. Fam Plann Perspect. 1998 Nov-Dec;30(6):271-5. PMID 9859017
- [Background] DiClemente RJ, Crosby RA, Wingood GM, Lang DL, Salazar LF, Broadwell SD. Reducing risk exposures to zero and not having multiple partners: findings that inform evidence-based practices designed to prevent STD acquisition. Int J STD AIDS. 2005 Dec;16(12):816-8. doi: 10.1258/095646205774988037. PMID 16336765
- [Background] Muzny CA, Austin EL, Harbison HS, Hook EW 3rd. Sexual partnership characteristics of African American women who have sex with women; impact on sexually transmitted infection risk. Sex Transm Dis. 2014 Oct;41(10):611-7. doi: 10.1097/OLQ.0000000000000194. PMID 25211257
- [Background] Muzny CA, Harbison HS, Austin EL, Schwebke JR, Van Der Pol B, Hook EW 3rd. Sexually Transmitted Infection Risk among Women Is Not Fully Explained by Partner Numbers. South Med J. 2017 Mar;110(3):161-167. doi: 10.14423/SMJ.0000000000000621. PMID 28257539